CLINICAL TRIAL: NCT04116450
Title: Microcatheter Assisted Circumferential Trabeculotomy in Congenital Glaucoma
Brief Title: MicrocatheterTrabeculotomy in Primary Congenital Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Shaaban Elwan, Assistant professor of ophthalmology, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Minia U, Glaucoma unit
Record Dates: First submitted 2019-10-01; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Primary Congenital Glaucoma
MeSH Terms: conditions — Hydrophthalmos

STUDY DESIGN:
Intervention Model Description: 25 patient underwent Glaucolight illuminated microcatheter for primary congenital glaucoma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- primary congenital glaucoma (Other): Glaucolight illuminated microcatheter trabeculotomy in primary congenital glaucoma
  Interventions: Procedure: Glaucolight illuminated microcatheter.

INTERVENTIONS:
Procedure: Glaucolight illuminated microcatheter. — To study circumferential trabeculotomy for congenital glaucoma using Glaucolight illuminated microcatheter.
  Other Names: circumferential trabeculotomy for congenital glaucoma using Glaucolight illuminated microcatheter.

SUMMARY:
PURPOSE: To study circumferential trabeculotomy for congenital glaucoma using Glaucolight illuminated microcatheter.

Setting: Ophthalmology department, Faculty of Medicine, Minia University, 61519, El-Minia, Egypt.

DESIGN: Prospective, randomized, consecutive interventional study

METHODS:

This was a prorospective study of 25 eyes of 25 patients with primary congenital or juvenile glaucoma those underwent circumferential trabeculotomy done with an illuminated microcatheter through a period of 24 months. Patients data of 12 months follow-up were recorded. The primary target was mean intraocular pressure (IOP) study in which unqualified (complete success) was defined as an IOP ≤21 mm Hg and at least a 30% reduction without the use of antiglaucoma drugs and a qualified success when medications were used to reach this aim. The secondary target was studding the corneal diameter (CD) and cup disc ratio (C/D) change.

DETAILED DESCRIPTION:
Subjects and Methods This was a prorospective study of 25 eyes of 25 patients with primary congenital or juvenile glaucoma those underwent circumferential 360° trabeculotomy done with an illuminated microcatheter (DORC International, Zuidland, Netherlands) through a period of 24 months from June 2017 to May 2019. The child parents were informed by the procedure and signed a consent as well as the study was approved from Ethical Committees and was in accordance with the Declaration of Helsinki.

inclusion criteria: The study included children aged below 6 years with PCG with or without antiglaucoma medications and not had previous antiglaucoma surgery with successful 360°trabeculotomy.

Exclusion criteria: Eyes that needs combined operation, previous antiglaucoma procedure and incomplete trabeculotomy ≤360°.

Preoperative examinations: Routine ocular examination or under general anesthesia for younger children were done after history taking including, age, sex, laterality, family history and consanguinity, antiglaucoma drugs. The ocular examinations includes IOP with Goldman applanation or Perkins tonometer, slit lamp, corneal clarity, measurement of horizontal corneal diameter, axial length by ultrasonography and fundus examination and measurement of cup disc ratio. The demographic data were registered as in (Table 1).

Surgical procedure:

Under general anesthesia, routine ophthalmology srcupping and sterilization. Eye speculum was inserted then

* Conjunctival peritomy with fornix based flap was done.
* Superficial rectangular scleral flab 3.5 x 4.5 mm and deep scleral flab 2 x 3 mm with deroofing of Sclemm's canal anteriorly to the scleral spur were done.
* Cutting Sclemm's canal and exposure of its ostia and dilatation of the ostia by injection of Healon.
* Paracentesis to lower IOP and injection of Miochol for miosis and Healon to keep anterior chamber stable and deep.
* Introducing the illuminated catheter into one of the Sclemm's canal ostium and advanced through the whole Sclemm's canal 360° circumference.
* When the atraumatic tip of the catheter appeared from the other ostium, both ends were pulled in opposite direction to make 360° trabeculotomy.
* Both Scleral flaps were closed with interrupted 10/0 nylon suture and Conjunctival flap with contentious 10/0 nylon suture.
* Injection of subconjunctival steroid and antibiotic, then eye dressing.

Post-operative management :

The patients were prescribed topical tobradex( tobramycin- dexamethasone) eye drops QID and tapering through 4-6 weeks and topical cycloplegic eye drops TID for 3 days. Scheduled follow up visits were advised next postoperative day, one week, monthly for three months then each three months till one year. Each visit the child subjected to full ophthalmological examinations previously mentioned and antiglaucoma medications were prescribed when needed (IOP<21 mmHg) or appearing of signs of glaucoma progression starting by one drug beta blockers and adding dorzolamide or prostaglandin to reach the target IOP.

Patients data of 12 months follow-up were recorded. The primary target was mean intraocular pressure (IOP) study in which unqualified (complete success) was defined as an IOP ≤21 mm Hg and at least a 30% reduction without the use of antiglaucoma drugs, a qualified success when medications were used to reach this aim and failure if the target IOP would not reached in spite of full antiglaucoma medication and the child needs another antiglaucoma procedure. The secondary target was studding the corneal diameter (CD) and cup disc ratio (C/D) change. The results of one week, 3 months, 6 months and one year were included in the statistical analysis.

statistical analysis: Data were collected, revised, verified, coded, then entered PC for statistical analysis done by using SPSS statistical package version 20. Descriptive statistics for quantitative data: mean (X) and standard deviation (SD). Kolmogorov- Smirnov for normality test was used to differentiate between parametric data and non-parametric data. Statistical analysis using Wilcoxon signed ranks test for comparison of two related parameters preoperative and postoperative. For all tests probability (P value) was considered non-significant if ≥ 0.05, significant if < 0.05, highly significant if < 0.01 and very highly significant if <0.001.

ELIGIBILITY:
Inclusion Criteria:

* The study included children aged below 6 years with PCG with or without antiglaucoma medications and not had previous antiglaucoma surgery with successful 360°trabeculotomy.

Exclusion Criteria:

* Eyes that needs combined operation, previous antiglaucoma procedure and incomplete trabeculotomy ≤360°.

Ages: 2 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Intra-ocular pressure | one year
  The primary target was mean intraocular pressure (IOP) study in which unqualified (complete success) was defined as an IOP ≤21 mm Hg and at least a 30% reduction without the use of antiglaucoma drugs and a qualified success when medications were used to reach this aim.

SECONDARY OUTCOMES:
corneal diameer | 1 year
  The secondary target was studding the corneal diameter (CD)
cup discratio | 1 year
  cup disc ratio (C/D) change.

CONTACTS AND LOCATIONS:
Overall Officials: mahmoud M Genaidy, MD, Study Director — Minia University
Locations (1):
- Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No
freely share

REFERENCES:
- [Background] El Sayed Y, Gawdat G. Two-year results of microcatheter-assisted trabeculotomy in paediatric glaucoma: a randomized controlled study. Acta Ophthalmol. 2017 Dec;95(8):e713-e719. doi: 10.1111/aos.13414. Epub 2017 Mar 7. PMID 28266150
- [Background] Morales J, Al Shahwan S, Al Odhayb S, Al Jadaan I, Edward DP. Current surgical options for the management of pediatric glaucoma. J Ophthalmol. 2013;2013:763735. doi: 10.1155/2013/763735. Epub 2013 Apr 24. PMID 23738051